CLINICAL TRIAL: NCT04656132
Title: Physical Activity Assessment, Promotion and Monitoring in a Preventive Cardiology Clinic: A Pilot Study
Brief Title: PAVS in Cardiology
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-00388
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with cardiovascular disease or cardiovascular disease risk factors (Experimental): Population We will recruit 59 males and females age > 18 being seen in the NYU Langone Center for Prevention of Cardiovascular Disease (4F). Participants have cardiovascular disease or cardiovascular disease risk factors.
  Interventions: Behavioral: Physical activity assessment, promotion and monitoring in a preventive cardiology clinic

INTERVENTIONS:
Behavioral: Physical activity assessment, promotion and monitoring in a preventive cardiology clinic — physical activity assessment promotion and remote home step-count monitoring in a clinical cardiology center

SUMMARY:
Brief Summary This is a pilot study implemented physical activity assessment, promotion and monitoring in patients. Patients will be assessed by the physical activity vital sign (PAVS) during check-in for their appointment. During their visit with the cardiologist, a clinical decision support tool will alert the cardiologist to patients achieving low (<50% of recommended) physical activity. The cardiologist may refer the patient to cardiac rehabilitation if appropriate and/or counsel them to increase their physical activity levels. The patients may opt to enroll in the monitoring phase of the study. They will be given a Fitbit pedometer and their Fitbit account can sync to their MyChart account. After that sync, the patients step counts will be available for their cardiologists to review as needed.

ELIGIBILITY:
Inclusion Criteria:

Adult patients in the Center who are age 18 and above will be assessed with the PAVS as part of routine care. To enroll in the home monitoring of PA:

1. Patients must achieve < 50% of PA recommendations according to PAVS screening questions
2. Have a cellular phone with data plan or a computer to sync Fitbit data
3. Speak English or Spanish
4. Be willing to wear a Fitbit Zip for 3 months

Exclusion Criteria:

1. Adults with a physical disability or medical diagnosis limiting their ability to exercise (e.g. wheelchair bound, aortic stenosis, unstable angina)
2. Planned surgery within three months
3. Those with decisional incapacity therefore unable to comply with study requirements (i.e. related to cognitive deficits or psychiatric diagnosis)
4. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Langone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to:mmm529@nyu.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 months and ending 36 months following article publication
Access Criteria: Requests should be directed to mmm529@nyu.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] McCarthy MM, Szerencsy A, Taza-Rocano L, Hopkins S, Mann D, D'Eramo Melkus G, Vorderstrasse A, Katz SD. Implementing a Clinical Decision Support Tool to Improve Physical Activity. Nurs Res. 2024 May-Jun 01;73(3):216-223. doi: 10.1097/NNR.0000000000000714. Epub 2024 Jan 11. PMID 38207172

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Cardiovascular Disease or Cardiovascular Disease Risk Factors
Started | 63
Completed | 55
Not Completed | 8
Not completed — Lost to Follow-up | 4
Not completed — Lost to Follow-Up Prior to Baseline Data Collection | 4

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Cardiovascular Disease or Cardiovascular Disease Risk Factors
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.13 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 45
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Step Counts
Description: Pedometer
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Participants With Cardiovascular Disease or Cardiovascular Disease Risk Factors
Number analyzed (Participants) | 55
steps | 48770 (27362)

2. Primary Outcome: BMI
Description: BMI will be calculated by height and weight measured at the time of the Center visit on a balance beam scale.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Participants With Cardiovascular Disease or Cardiovascular Disease Risk Factors
Number analyzed (Participants) | 55
kg/m^2 | 30 (7)

3. Primary Outcome: Waist Circumference
Description: Waist Circumference will be measured to the nearest inch using standard technique
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Participants With Cardiovascular Disease or Cardiovascular Disease Risk Factors
Number analyzed (Participants) | 55
inches | 38.9 (6)

4. Primary Outcome: Blood Pressure
Description: Blood pressure (BP) will be measured in right arm (unless contraindicated) after sitting for 5 minutes and repeated after a 5-minute interval. Both will be recorded and the average used in analyses.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Participants With Cardiovascular Disease or Cardiovascular Disease Risk Factors
Number analyzed (Participants) | 55
mmHg
  Systolic | 125 (16)
  Diastolic | 76 (14)

5. Primary Outcome: Blood Lipid Levels
Description: Total cholesterol, HDL, and triglycerides will be measured by CLIA-waived Alere Cholestech LDX® Analyzer which is certified by the Center for Disease Control's Lipid Standardization Program and Cholesterol Reference Method Laboratory Method Network. This will be measured by a single fingerstick using standard aseptic technique.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Participants With Cardiovascular Disease or Cardiovascular Disease Risk Factors
Number analyzed (Participants) | 55
mg/dl
  Cholesterol | 148 (45)
  HDL | 43 (18)
  Triglycerides | 138 (76)

6. Primary Outcome: Framingham Heart Study Risk Score
Description: The Framingham Heart Study Risk Score (10-year risk) will be calculated using the appropriate risk model based on participants' age, gender, diabetes status and prior coronary heart disease. Risk is considered low if the FRS is less than 10%, moderate if it is 10% to 19%, and high if it is 20% or higher.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: Percentage risk
Arm/Group | Participants With Cardiovascular Disease or Cardiovascular Disease Risk Factors
Number analyzed (Participants) | 55
Percentage risk | 8.6 (9.7)

ADVERSE EVENTS:
Time Frame: 3 months
Description: PI monitored for adverse events systematically at the followup visit, and informally during the study period with self-reporting by the subjects.
Arm/Group | Participants With Cardiovascular Disease or Cardiovascular Disease Risk Factors
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 1/63
Other Adverse Events (participants affected / at risk) | 1/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Cardiovascular Disease or Cardiovascular Disease Risk Factors (N=63)
Hospitalization for an Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Cardiovascular Disease or Cardiovascular Disease Risk Factors (N=63)
Hip Fracture (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT04656132/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT04656132/ICF_002.pdf